CLINICAL TRIAL: NCT05479253
Title: A Single-center Study of an AI-assisted Endoscopy Report System In Improving Reporting Quality
Brief Title: AI-assisted Endoscopy Report System In Improving Reporting Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: EA-21-010
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-07

CONDITIONS: Artificial Intelligence; Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with Artificial intelligence assistant system (Experimental): Endoscopists would complete the endoscopy report with the assistance of the artificial intelligence system.
  Interventions: Diagnostic Test: Artificial intelligence assistant system
- without Artificial intelligence assistant system (No Intervention): Endoscopists would complete the endoscopy report without special prompts.

INTERVENTIONS:
Diagnostic Test: Artificial intelligence assistant system — The artificial intelligence assistant system can automatically capture images, prompt abnormal lesions and the parts covered by the examination (the stomach is divided into 26 parts).
  Arms: with Artificial intelligence assistant system

SUMMARY:
In this study, we proposed a prospective study about the effectiveness of artificial intelligence system for endoscopy report quality in endoscopists. The subjects would be divided into two groups. For the collected endoscopic videos, group A would complete the endoscopy report with the assistance of the artificial intelligence system. The artificial intelligence assistant system can automatically capture images, prompt abnormal lesions and the parts covered by the examination (the upper gastrointestinal tract is divided into 26 parts). Group B would complete the endoscopy report without special prompts. After a period of forgetting, the two groups switched, that is, group A without AI assistance and group B with AI assistance to complete the endoscopy report. Then, the completeness of the report lesion, the accuracy of the lesion location, the completeness of the lesion and the standard part in the captured images, and so on were compared with or without AI assistance.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females who are over 18 years old;
2. After qualified medical education and obtained the Certificate of Chinese medical practitioner;

Exclusion Criteria:

1. Doctors without qualified medical education and didn't obtaine the Certificate of Chinese medical practitioner;
2. The researcher believes that the subjects are not suitable for participating in clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Integrity of report lesion | one month
  Report lesion integrity with or without AI-assisted. Calculation method = number of report lesions / total number of lesions x 100%
Accuracy of lesion location | one month
  Accuracy of lesion location with or without AI-assisted. Calculation method = number of lesion with correct location / total number of lesions x 100%
Integrity of lesion in captured images | one month
  Lesion integrity in captured images with or without AI-assisted. Calculation method = number of lesions in captured images / total number of lesions x 100%
Integrity of standard part in captured images | one month
  Lesion integrity in captured images with or without AI-assisted. Calculation method = number of standard parts in captured images / the actual number of standard parts covered by the examination x 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Lu Z, Yao L, Dong Z, Zhou W, He C, Luo R, Zhang M, Wang J, Li Y, Deng Y, Zhang C, Li X, Shang R, Xu M, Wang J, Zhao Y, Wu L, Yu H. Effect of a deep learning-based automatic upper GI endoscopic reporting system: a randomized crossover study (with video). Gastrointest Endosc. 2023 Aug;98(2):181-190.e10. doi: 10.1016/j.gie.2023.02.025. Epub 2023 Feb 25. PMID 36849056